CLINICAL TRIAL: NCT03922165
Title: Healthy Sleep for Children With Down Syndrome
Acronym: HELP-DS
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University Hospitals Cleveland Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Michigan (Other); University of Texas Southwestern Medical Center (Other); University of Rochester (Other); Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, Susan Redline, Professor, Brigham and Women's Hospital
Other Study IDs: 18-015848
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Down Syndrome; Sleep Disordered Breathing
Keywords: Pediatrics; Adenotonsillectomy
MeSH Terms: conditions — Down Syndrome; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DS peds eligible for Adenotonsillectomy: Dyads of caregivers and children with DS aged 3-13 years diagnosed with SDB and referred for treatment with adenotonsillectomy.
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Adenotonsillectomy — Routine AT per clinical care.

SUMMARY:
The purpose of this multi-center observational study (utilizing the sites enrolling patients for the Pediatric Adenotonsillectomy Trial for Snoring (PATS) [1U011HL125307-O1A1]) is to gather data regarding children with Down syndrome (DS) and Sleep Disordered Breathing (SDB) referred for treatment with adenotonsillectomy to inform a future randomized controlled trial in this population.

DETAILED DESCRIPTION:
Down syndrome (DS) is associated with a wide range of neurobehavioral and physical morbidities. Obstructive sleep apnea (OSA) is prevalent in children with DS and causes a myriad of physiological stresses that may exacerbate neurobehavioral and cardiac morbidities. Improving sleep health thus provides a modifiable intervention target for improving behavior, cognition, quality of life, and physical health of children with DS. However, critical knowledge gaps limit the adoption and implementation of effective OSA interventions, resulting in practice variability and suboptimal treatment of OSA across the spectrum of DS. In particular, it is in unclear how to select candidates likely to benefit from adenotonsillectomy (AT) and how to utilize information from polysomnographic, clinical, and demographic parameters to predict children most likely to benefit from AT compared to alternative treatments or to watchful waiting. The goal of this study is to collect the necessary data to plan and execute a future pivotal RCT of the role of OSA treatment in the care of children with DS. This study will provide critical information on the methodological approaches for conducting such a randomized controlled clinical trial (RCT), informing the appropriate recruitment strategies, patient population and outcome measures for a future clinical trial. The investigators will leverage expertise in pediatric sleep medicine, clinical trials, neuropsychology, and DS as well as the PATS clinical trials infrastructure to catalyze a new DS clinical research initiative. Our proposed next steps are to enroll in an observational study at active PATS centers 50 children with DS who are referred for clinically indicated evaluation and treatment of OSA. At baseline and 6 months following AT, these children will undergo systematic assessments of sleep, behavior, cognition, daytime functioning, and quality of life, generating key data to inform the design of a later pivotal RCT.

Healthy Sleep for Children with Down Syndrome (HELP-DS) intends to take advantage of a successful collaboration of leaders in sleep medicine, otolaryngology and clinical trials to efficiently leverage experiences from the The Childhood Adenotonsillectomy Trial (CHAT) as well as the current resources of the PATS trial to collect data for the evaluation of key questions needed to design a future RCT, including approaches related to the selection of participating sites, the patient population to receive the intervention, and outcome measurements.

The primary objective of HELP-DS to determine the feasibility of recruiting and retaining individuals in an observational study of AT across multiple clinical sites.

Secondary objectives are:

1. Evaluate the feasibility of collecting a range of baseline and outcome data, and specifically the ability of children to perform neurobehavioral assessments (GoNoGo, pegboard task).
2. Understand issues related to patient preference, equipoise, and barriers to treatment. The investigators will track how many children referred for AT actually undergo surgery, the time interval between referral and surgery, other interventions pursued, and factors such as insurance, socio-economic factors, and cultural norms, that associate with family-decision making.
3. Examine the consistency and completeness of Healthcare Utilization (HCU) data extracted across our sites, describing differences by recruitment site, health, system characteristics, insurance-related factors, etc. The investigators will estimate incidence rates of HCU events for hospital admissions, emergency department/unscheduled office visits, specialty consultations and medication use during the 6 months following surgery and compare rates to those for the year prior to surgery.

These aims have substantial public health significance given the high morbidity of Down syndrome and sleep-disordered breathing in children.

ELIGIBILITY:
Inclusion Criteria:

* DS diagnosis regardless of genetic status (e.g., mosaicism or translocation).
* Aged >3 to <13 years at the date of consent.
* Primary indication for AT is nocturnal obstructive symptoms (i.e., not recurrent infections or other indications).
* Deemed to be a candidate for AT by Ear, Nose and Throat (ENT) evaluation; that is, no technical issues that would be a contraindication for surgery such as submucous cleft palate.

Exclusion Criteria:

* Prior tonsillectomy (partial or complete).
* Severe chronic health conditions that would contradict surgery (severe morbid obesity, unrepaired cyanotic congenital heart disease, bleeding disorders).
* Severe behavioral problems that would preclude participation in the study's testing procedures (PSG, actigraphy).
* Severe OSA with respiratory failure needing urgent/emergent management
* Plan to undergo additional airway surgery at the time of AT.
* Caregiver/child planning to move out of the area within 6 months.
* Caregiver/child does not speak English or Spanish well enough to complete the behavioral and performance measures.
* Child in foster care.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Dyads of caregivers and children with DS aged 3-13 years diagnosed with SDB and referred for treatment with adenotonsillectomy (AT) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
% enrolled/approached | 1 year
  Percentage of families approached for participation that sign informed consent to participate.
% retained/enrolled | 1 year
  Percentage of consented families that completed study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Rui Wang, PhD, Principal Investigator — Brigham and Women's Hospital; Susan L Furth, Md, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals-Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia

REFERENCES:
- [Background] Mai CT, Kucik JE, Isenburg J, Feldkamp ML, Marengo LK, Bugenske EM, Thorpe PG, Jackson JM, Correa A, Rickard R, Alverson CJ, Kirby RS; National Birth Defects Prevention Network. Selected birth defects data from population-based birth defects surveillance programs in the United States, 2006 to 2010: featuring trisomy conditions. Birth Defects Res A Clin Mol Teratol. 2013 Nov;97(11):709-25. doi: 10.1002/bdra.23198. No abstract available. PMID 24265125
- [Background] Presson AP, Partyka G, Jensen KM, Devine OJ, Rasmussen SA, McCabe LL, McCabe ER. Current estimate of Down Syndrome population prevalence in the United States. J Pediatr. 2013 Oct;163(4):1163-8. doi: 10.1016/j.jpeds.2013.06.013. Epub 2013 Jul 23. PMID 23885965
- [Background] Sherman SL, Allen EG, Bean LH, Freeman SB. Epidemiology of Down syndrome. Ment Retard Dev Disabil Res Rev. 2007;13(3):221-7. doi: 10.1002/mrdd.20157. PMID 17910090
- [Background] Bull MJ; Committee on Genetics. Health supervision for children with Down syndrome. Pediatrics. 2011 Aug;128(2):393-406. doi: 10.1542/peds.2011-1605. Epub 2011 Jul 25. PMID 21788214
- [Background] Yang Q, Rasmussen SA, Friedman JM. Mortality associated with Down's syndrome in the USA from 1983 to 1997: a population-based study. Lancet. 2002 Mar 23;359(9311):1019-25. doi: 10.1016/s0140-6736(02)08092-3. PMID 11937181
- [Background] Rajagopal KR, Abbrecht PH, Derderian SS, Pickett C, Hofeldt F, Tellis CJ, Zwillich CW. Obstructive sleep apnea in hypothyroidism. Ann Intern Med. 1984 Oct;101(4):491-4. doi: 10.7326/0003-4819-101-4-491. PMID 6476635
- [Background] Marcus CL, Keens TG, Bautista DB, von Pechmann WS, Ward SL. Obstructive sleep apnea in children with Down syndrome. Pediatrics. 1991 Jul;88(1):132-9. PMID 1829151
- [Background] de Miguel-Diez J, Villa-Asensi JR, Alvarez-Sala JL. Prevalence of sleep-disordered breathing in children with Down syndrome: polygraphic findings in 108 children. Sleep. 2003 Dec 15;26(8):1006-9. doi: 10.1093/sleep/26.8.1006. PMID 14746382
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Edgin JO, Tooley U, Demara B, Nyhuis C, Anand P, Spano G. Sleep Disturbance and Expressive Language Development in Preschool-Age Children With Down Syndrome. Child Dev. 2015 Nov-Dec;86(6):1984-98. doi: 10.1111/cdev.12443. Epub 2015 Oct 5. PMID 26435268
- [Background] Clausen J, Sersen EA, Lidsky A. Sleep patterns in mental retardation: Down's syndrome. Electroencephalogr Clin Neurophysiol. 1977 Aug;43(2):183-91. doi: 10.1016/0013-4694(77)90126-2. PMID 69529
- [Background] Nisbet LC, Phillips NN, Hoban TF, O'Brien LM. Characterization of a sleep architectural phenotype in children with Down syndrome. Sleep Breath. 2015 Sep;19(3):1065-71. doi: 10.1007/s11325-014-1094-6. Epub 2014 Dec 12. PMID 25500979
- [Background] Diomedi M, Curatolo P, Scalise A, Placidi F, Caretto F, Gigli GL. Sleep abnormalities in mentally retarded autistic subjects: Down's syndrome with mental retardation and normal subjects. Brain Dev. 1999 Dec;21(8):548-53. doi: 10.1016/s0387-7604(99)00077-7. PMID 10598057
- [Background] Reckley LK, Fernandez-Salvador C, Camacho M. The effect of tonsillectomy on obstructive sleep apnea: an overview of systematic reviews. Nat Sci Sleep. 2018 Apr 4;10:105-110. doi: 10.2147/NSS.S127816. eCollection 2018. PMID 29670412
- [Background] Farhood Z, Isley JW, Ong AA, Nguyen SA, Camilon TJ, LaRosa AC, White DR. Adenotonsillectomy outcomes in patients with Down syndrome and obstructive sleep apnea. Laryngoscope. 2017 Jun;127(6):1465-1470. doi: 10.1002/lary.26398. Epub 2017 Jan 5. PMID 28055122
- [Background] Garetz SL, Mitchell RB, Parker PD, Moore RH, Rosen CL, Giordani B, Muzumdar H, Paruthi S, Elden L, Willging P, Beebe DW, Marcus CL, Chervin RD, Redline S. Quality of life and obstructive sleep apnea symptoms after pediatric adenotonsillectomy. Pediatrics. 2015 Feb;135(2):e477-86. doi: 10.1542/peds.2014-0620. Epub 2015 Jan 19. PMID 25601979
- [Background] Franco RA Jr, Rosenfeld RM, Rao M. First place--resident clinical science award 1999. Quality of life for children with obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):9-16. doi: 10.1067/mhn.2000.105254. PMID 10889473
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Arozullah AM, Yarnold PR, Bennett CL, Soltysik RC, Wolf MS, Ferreira RM, Lee SY, Costello S, Shakir A, Denwood C, Bryant FB, Davis T. Development and validation of a short-form, rapid estimate of adult literacy in medicine. Med Care. 2007 Nov;45(11):1026-33. doi: 10.1097/MLR.0b013e3180616c1b. PMID 18049342
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376